CLINICAL TRIAL: NCT06317480
Title: Does Composite Bone Resection for Soft Tissue Sarcoma With Cortical Contact Result in Better Local Control and Survival Compared to Sub-periosteal Dissection?
Brief Title: Outcomes Comparison Between Bone Resection and Subperiosteal Dissection for Specific Type of Soft Tissue Sarcoma
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: QH_2024
Record Dates: First submitted 2024-03-04; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Soft Tissue Sarcoma; Cortical Contact
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bone resection
  Interventions: Procedure: bone resection
- subperiosteal excision
  Interventions: Procedure: subperiosteal excision

INTERVENTIONS:
Procedure: bone resection — patients underwent soft tissue sarcoma excision together with bone resection following either biological or endoprosthesis reconstruction
  Groups: bone resection
Procedure: subperiosteal excision — patients underwent sub-periosteal tumor excision combining bone and soft tissue ablation without bone excision
  Groups: subperiosteal excision

SUMMARY:
the purpose of this study is to assess whether bone resection for thigh soft tissue sarcoma with cortical involvement of the adjacent bone result in better local control and survival compared to sub-periosteal dissection. Investigators also aim to find out the prognostic factors for clinical outcomes in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients developed thigh soft tissue sarcoma, defined as lesion located below the plane of the lesser trochanter and above the plane of the femoral condyle.
2. received primary limb-salvage surgery at our center.
3. soft tissue sarcoma with only cortical contact of the adjacent bone based on preoperative imaging
4. minimum of 2-year follow up

Exclusion Criteria:

1. diagnosis was well differentiated liposarcoma
2. patients with metastatic disease at the time of presentation
3. soft tissue sarcoma displayed frank osseous invasion (eg. medullary canal invasion)

Ages: 8 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients displayed with thigh soft tissue sarcoma with only cortical contact of the adjacent bone and underwent limb-salvage surgery were included for the study. Patients could be divided into two groups: 1) sub-periosteal tumor excision group and 2) composite bone resection and reconstruction group.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2000-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
survival | patients were checked every three months for the initial two years after surgery and every 6 months for the subsequent three years. After 5 years, patients will be checked once every year until patients died or were loss to follow up.
  Whether patient die or not
recurrence | patients were checked every three months for the initial two years after surgery and every 6 months for the subsequent three years. After 5 years, patients will be checked once every year until patients died or were oss to follow up.
  whether patients developed local recurrence
metastasis | patients were checked every three months for the initial two years after surgery and every 6 months for the subsequent three years. After 5 years, patients will be checked once every year until they died or were loss to follow up.
  whether patients developed metastasis

SECONDARY OUTCOMES:
functional outcomes | MSTS scores were measured every 6 months for the first two years after surgery. After that, MSTS outcomes were measured once every year until patients died or were loss to follow up.
  The Musculoskeletal Tumor Society (MSTS) questionnaire for the lower extremity is composed of six items including pain, function, emotional acceptance, use of any external support, walking ability, and gait alteration. Each item is rated in a scale of 0-5. The total score ranges from 0 to 30, with higher scores indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoming Ye, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: No